CLINICAL TRIAL: NCT01487811
Title: Bioequivalence of Two Biphasic Insulin Aspart 30 (NovoLog® Mix 70/30) Formulations (Current and New Formulation With Glycerol): A Randomized, Double-Blind, Two-Period Crossover Study in Healthy Volunteers
Brief Title: Comparison of Two Biphasic Insulin Aspart 30 Formulations (Current and New Formulation) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1669
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation 1 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30
- Formulation 2 (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Single dose administrated subcutaneously (s.c., under the skin)

SUMMARY:
This trial is conducted in the United states of America (USA). The aim of this trial is to compare two formulations of biphasic insulin aspart 30 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* BMI (body mass index) between 18 and 28 kg/m^2, both inclusive
* Subject is a nonsmoker for at least 3 months
* Subject is judged to be in good health on the basis of their medical history, physical examination, ECG (electrocardiogram), and routine laboratory data
* Fasting plasma glucose between 80 and 110 mg/dl

Exclusion Criteria:

* •Any clinically significant disease history of systemic or organ disease
* •Clinically significant abnormalities on pre-study clinical examination or any laboratory measurements during screening (any abnormality should be discussed with the clinical monitor)
* •In females of child bearing potential: Pregnancy, lactating, breastfeeding, intent to become pregnant within the next 6-months or judged to be using inadequate contraceptive measures (adequate contraceptive measures include: condom, intrauterine devices). ß-hCG pregnancy test must be negative

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2005-05; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Area under the concentration curve (AUC) of the two formulations from time 0 hours to infinity
Maximum drug concentration of the two formulations (Cmax)

SECONDARY OUTCOMES:
Area under the concentration curve for insulin aspart from time 0 hours to 16 hours
Mean residence time (MRT)
Frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, San Antonio, Texas, United States

REFERENCES:
- [Result] Hanefeld M, Fischer S, Julius U, Schulze J, Schwanebeck U, Schmechel H, Ziegelasch HJ, Lindner J. Risk factors for myocardial infarction and death in newly detected NIDDM: the Diabetes Intervention Study, 11-year follow-up. Diabetologia. 1996 Dec;39(12):1577-83. doi: 10.1007/s001250050617. PMID 8960845
- [Result] Standl E, Balletshofer B, Dahl B, Weichenhain B, Stiegler H, Hormann A, Holle R. Predictors of 10-year macrovascular and overall mortality in patients with NIDDM: the Munich General Practitioner Project. Diabetologia. 1996 Dec;39(12):1540-5. doi: 10.1007/s001250050612. PMID 8960840
- [Result] The absence of a glycemic threshold for the development of long-term complications: the perspective of the Diabetes Control and Complications Trial. Diabetes. 1996 Oct;45(10):1289-98. PMID 8826962
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com